CLINICAL TRIAL: NCT01402570
Title: Oral Glutathione and Health Outcomes Among Persons With Post-Polio Syndrome
Brief Title: Glutathione and Health With Post-Polio Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Claire Z. Kalpakjian, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPH-1051
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Post-polio Syndrome; Physical Activity; Depression; Pain; Sleep Disorders
Keywords: disability; polio; rehabilitation; wellness
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Motor Activity; Depression; Pain; Sleep Wake Disorders; Poliomyelitis | interventions — Glutathione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glutathione supplement (Experimental): All subjects will be taking a glutathione supplement.Glutathione is a naturally occuring antioxidant and a nonessential amino acid.
  Interventions: Dietary Supplement: Glutathione

INTERVENTIONS:
Dietary Supplement: Glutathione — glutathione is a dietary supplement and an antioxidant. Subjects will take 1000 mg per day for three month. Each capsule contains 500 mg glutathione.
  Other Names: 500 Ultrathoine, GSH and l-glutathione.

SUMMARY:
In this study, people who have symptoms of post polio will take oral glutathione supplements for three months. Their levels of fatigue, physical activity and sleep efficiency will be assessed.

DETAILED DESCRIPTION:
Subjects will take a glutathione supplement by mouth for three months after an initial medical visit, blood draw and physical exam. There are four timepoints during the three months when subjects will fill out surveys and record food intake and sleep times in diaries for seven days. They will also wear a small device for seven days, a Sensewear monitor that records physical activity, body temperature and other measures.

After the fourth timepoint they will return to the medical center for another physical exam and blood draw. Physicians trained in physical medicine and rehabilitation will be monitoring the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk 100 feet with usual assistive devices (ex. cane or walker)
* Having a function score of 18-32 when tested with the IPPS (Index of Post- Polio Sequelae). This will include people with post-polio symptoms in a very specific range of severity.

Exclusion Criteria:

* Having another serious medical condition (cancer, multiple sclerosis, etc.)or inflammatory disease (ie., lupus)
* Currently taking glutathione or other antioxidants

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Kalpakjian, PhD, MS, Principal Investigator — University of Michigan; Mark Ziadeh, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: All subjects took a three month trials of 1,000 mg of glutathione supplement
Period: Overall Study
Arm/Group | Study Group
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The target population for this study was individuals between the ages of 50 and 65 who self-reported symptoms consistent with post-polio syndrome and able to ambulate 100 feet without assistive devices.
Groups:
- Study Group: All subjects were assigned the intervention. The intervention was a three-month trial of twice daily, oral, 1,000 mg glutathione supplements (Glutathione 500 Ultrathione, The Glutathione Corporation, Elmsford, New York; 500 mg. capsule with 250 mg. ascorbic acid).
Arm/Group | Study Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.85 (3.89)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
PROMIS Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — Assesses the ability to carry out activities that require physical actions, ranging from self-care (activities of daily living) to more complex activities that require a combination of skills, often within a social context. Scores are standardized T-scores with mean of 50 and standard deviation of 10; higher scores indicate better physical function.
  units on a scale | 37.8 (4.6)
Subjective sleep efficiency [Mean (Standard Deviation); unit: percentage] — Sleep efficiency is defined as the ratio of time sleeping and time in bed. Using a sleep diary, participants recorded bedtime the night before, amount of time it took to fall asleep, number and total duration of awakenings, time of final awakening, and time of rising. Efficiency ranges from 0 to 100; higher values indicate higher sleep efficiency or more time sleeping when in bed.
  percentage | 82.0 (14.6)
PROMIS Fatigue [Mean (Standard Deviation); unit: units on a scale] — Assesses fatigue from mild subjective feelings to an overwhelming, debilitating, and sustained sense of exhaustion that is likely to decrease one's ability to carry out daily activities, including the ability to work effectively and to function at one's usual level in family or social roles. Fatigue is divided conceptually into the experience of fatigue (e.g., frequency, duration, and intensity), and the impact of fatigue upon physical, mental and social activities.Scores are standardized T-scores with mean of 50 and standard deviation of 10; higher scores indicate greater fatigue.
  units on a scale | 56.0 (8.7)
Physical activity, number of steps daily [Mean (Standard Deviation); unit: steps/day] — Refers to cumulative steps per day (24 hours period). 10,000 or more steps per day is considered optimal.
  steps/day | 4004.1 (3357.9)

OUTCOME MEASURES:

1. Primary Outcome: PROMIS (Patient Reported Outcomes Measurement Information System) Physical Functioning
Description: Ability to carry out activities that require physical actions, ranging from self-care (activities of daily living) to more complex activities that require a combination of skills, often within a social context. Scores are standardized T-scores with mean of 50 and standard deviation of 10; higher scores indicate better physical function.
Time Frame: Baseline, 1 month, 2 months and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 19
units on a scale
  Baseline | 37.8 (4.6)
  1 month | 37.9 (4.3)
  2 months | 37.5 (5.6)
  3 months | 38.1 (5.1)
Statistical Analysis 1: Comparison: Study Group; Linear mixed modeling (LMM) with random effects for intercept and repeated effects for assessment period was used to analyze change over time for study outcomes. The primary predictor of interest in this study was the relationship of time to each of the outcomes to evaluate the potential effect of the intervention. Independent LMMs were used to study outcomes; Test type: Superiority or Other; p = 0.66, Mixed Models Analysis — Time was predictor of interest, controlling for age, gender, baseline PROMIS physical functioning, and overall functional status; REML = 0.17, 95% CI 2-sided [-0.67 to 0.95]

2. Primary Outcome: Sleep Efficiency
Description: The ratio of time asleep over time in bed gathered from sleep diaries completed at bedtime and at awakening. Scores range from 0 to 100%, higher values indicate better sleep efficiency or more time sleeping in bed.
Time Frame: Baseline, 1 month, 2 months and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 19
units on a scale
  Baseline | 82.1 (14.6)
  1 month | 86.9 (9.2)
  2 months | 87.6 (8.4)
  3 months | 87.8 (8.2)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis — Time was predictor of interest, controlling for age, gender, baseline sleep efficiency, and overall functional status; REML = 0.00, 95% CI 2-sided [-0.01 to 0.02]

3. Primary Outcome: Steps Per Day
Description: Count of steps per day using activity monitor worn on upper arm.
Time Frame: Baseline, 1 month, 2 months and 3 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Study Group
Number analyzed (Participants) | 19
steps per day
  Baseline | 4004.1 (3357.9)
  1 month | 3590.7 (2928.3)
  2 months | 3598.9 (3139.3)
  3 months | 3693.1 (3317.8)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.35, Mixed Models Analysis — Time was predictor of interest, controlling for age, gender, baseline steps per day, and overall functional status; REML = 145.54, 95% CI 2-sided [-178.93 to 470.02]

4. Primary Outcome: PROMIS (Patient Reported Outcomes Measurement Information System) Fatigue
Description: Assesses fatigue from mild subjective feelings to an overwhelming, debilitating, and sustained sense of exhaustion that is likely to decrease one's ability to carry out daily activities, including the ability to work effectively and to function at one's usual level in family or social roles. Fatigue is divided conceptually into the experience of fatigue (e.g., frequency, duration, and intensity), and the impact of fatigue upon physical, mental and social activities. Scores are on a T-metric with mean of 50 and standard deviation of 10; higher scores indicate greater fatigue.
Time Frame: Baseline, 1 month, 2 months and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 19
units on a scale
  Baseline | 56.0 (8.7)
  1 month | 54.9 (7.1)
  2 months | 53.4 (9.2)
  3 months | 52.8 (9.8)
Statistical Analysis 1: Comparison: Study Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis — Time was predictor of interest, controlling for age, gender, baseline fatigue, and overall functional status; REML = -1.05, 95% CI 2-sided [-2.21 to 0.10]

ADVERSE EVENTS:
Time Frame: Entire study period of three months - baseline to the end of the trial.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=20)
allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size of 20 was quite small to make generalizations to the larger population. Dosing and duration of the intervention may not have been sufficient to effect change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No